CLINICAL TRIAL: NCT00369785
Title: Phase III Double Blind, Placebo Controlled Study of Donepezil in the Irradiated Brain
Brief Title: Donepezil in Treating Patients Who Have Undergone Radiation Therapy for Brain Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB00000551; U10CA081851 (NIH); REBACCCWFU 91105 (Other: NCI)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Brain Tumors; Metastatic Disease
Keywords: cognitive/functional effects; fatigue; psychosocial effects of cancer and its treatment; radiation toxicity; tumors metastatic to brain; adult brain stem glioma; adult central nervous system germ cell tumor; adult choroid plexus tumor; adult craniopharyngioma; adult mixed glioma; adult anaplastic meningioma; meningeal melanocytoma; adult meningeal hemangiopericytoma; adult grade I meningioma; adult grade II meningioma; adult grade III meningioma; adult papillary meningioma; adult anaplastic oligodendroglioma; adult oligodendroglioma; adult pineoblastoma; adult pineocytoma; adult anaplastic astrocytoma; adult diffuse astrocytoma; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma; adult pilocytic astrocytoma; adult ependymoblastoma; adult medulloblastoma; adult supratentorial primitive neuroectodermal tumor (PNET); adult anaplastic ependymoma; adult ependymoma; adult myxopapillary ependymoma; adult subependymoma
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis; Fatigue; Radiation Injuries; Choroid Plexus Neoplasms; Craniopharyngioma; Glioma; Meningioma; Oligodendroglioma; Pinealoma; Astrocytoma; Glioblastoma; Gliosarcoma; Neuroectodermal Tumors, Primitive; Medulloblastoma; Ependymoma; Glioma, Subependymal | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I - Donepezil (Experimental): Weeks 1-6: One 5 mg tablet orally donepezil hydrochloride Weeks 7-24: Two 5mg tablets per day
  Interventions: Drug: donepezil hydrochloride
- Arm II - Control (Placebo Comparator): Weeks 1-6: One placebo tablet per day Weeks 7-24: Two placebo tablets per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: donepezil hydrochloride — Weeks 1-6: One tablet Donepezil 5 mg given daily Weeks 7-24: Two Donepezil 5 mg tablets given daily
  Other Names: Donepezil
  Arms: Arm I - Donepezil
Drug: Placebo — Weeks 1-6: One tablet per day Weeks 7-24: Two tablets per day
  Arms: Arm II - Control

SUMMARY:
RATIONALE: Donepezil may help lessen confusion and fatigue and improve mood and quality of life in patients who have undergone radiation therapy for brain tumors. It is not yet known whether donepezil is more effective than a placebo in lessening side effects of radiation therapy in patients with brain tumors.

PURPOSE: This randomized phase III trial is studying donepezil to see how well it works in lessening side effects of radiation therapy compared with a placebo in patients who have undergone radiation therapy for brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effect of donepezil hydrochloride vs placebo, in terms of improving neurocognitive symptom cluster (i.e., cognitive impairment, subjective confusion, and fatigue), in patients who have undergone partial- or whole-brain irradiation for brain tumors.

Secondary

* Compare the effect of these regimens on mood and quality of life in these patients.

OUTLINE: This is a prospective, double-blind, placebo-controlled, randomized, multicenter study. Patients are stratified according to prior brain irradiation type (whole-brain vs partial-brain) and study site. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral donepezil hydrochloride once or twice daily for up to 24 weeks in the absence of unacceptable toxicity.
* Arm II: Patients receive oral placebo once or twice daily for up to 24 weeks in the absence of unacceptable toxicity.

Patients complete self-reported questionnaires (quality of life, fatigue, subjective confusion, neurocognitive battery, and mood) at baseline and 12 and 24 weeks.

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Adults >18 years old.
* Life expectancy of at least > 30 weeks.
* Must have received a prior course of at least 30 Gy fractionated whole or partial brain irradiation for treatment of a primary brain tumor or metastatic disease to the brain.
* Must have completed radiation > 6 months prior to enrollment and have no radiographic evidence of brain disease, or stable brain disease defined as no evidence of tumor progression in the 3 months prior to enrollment.
* Patients who have undergone one or more treatments with single fraction stereotactic radiosurgery (SRS) in addition to whole or partial brain irradiation are eligible, as long as the SRS was completed > 6 months prior to registration if NED or stable disease.
* Radiation treatment records must be available for all prior radiation treatments (external beam and/or SRS).
* Patients who have received PCI (prophylactic cranial irradiation) are eligible.
* Karnofsky Performance Status must be > 60 or ECOG 0-2.
* Treatment with steroids, anti-cholinergics, anti-epileptics, anti-depressants, and /or sedatives/benzodiazepines is acceptable, but the patient must be on a stable or decreasing dose at the time of study entry.
* Patients using narcotic analgesics on a stable dose and/or prn basis are eligible.
* Patients currently on a stable dose of Methylphenidate or Dextramphetamine are eligible.
* For patients with brain metastases, if extracranial primary or metastatic disease is present, it must have responded to local and/or systemic treatment. Must be stable in the 3 months prior to enrollment.
* Must not be receiving chemotherapy at the time of enrollment.
* Patient must not have any planned therapy, including surgery, brain radiation of any type, chemotherapy, or immunotherapy during the next 30 weeks for brain or extracranial primary metastatic disease.
* Hormonal therapy for patients with breast or prostate cancer is acceptable.
* Breast patients receiving therapy with Herceptin are allowed.
* Patients must be able to give informed consent to participate in the study, including signing the consent form.
* Patients must have a telephone.

EXCLUSION CRITERIA:

* Patients cannot be currently taking dementia drugs, cognitive enhancers, neuroleptics, and/or anti-parkinsonian agents. For patients who have used these drugs in the past, they must not have used them in the 2 weeks prior to enrolling on the study.
* Hypersensitivity to donepezil.
* Patients may not currently be taking Ketoconazole or Quindine
* Arrythmias including bradycardia or heartblock
* Patients who have received, GliaSite or other type of brain brachytherapy, (Gliadel Wafers permitted) convection enhanced delivery of immunotoxins, and/or any other investigational modalities for treatment of their brain tumor. The effects of donepezil on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* It is unknown whether donepezil is excreted in breast milk, for this reason women who are currently breast-feeding are not eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2012-07-01 (Actual); Study Completion 2012-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Rapp, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (16):
- United States (16):
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Central Maine Comprehensive Cancer Center at Central Maine Medical Center, Lewiston, Maine
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Trinity CancerCare Center, Minot, North Dakota
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Data Available: Select individual patient-level data form this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were accrued between 2/2008 and 12/2011 at NCI CCOP sites across the nation.
Period: Overall Study
Arm/Group | Arm I - Donepezil | Arm II - Control
Started | 99 | 99
Completed | 72 | 74
Not Completed | 27 | 25
Not completed — Physician Decision | 3 | 2
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Toxicity | 6 | 4
Not completed — Never started | 0 | 2
Not completed — Progression | 4 | 4
Not completed — Multiple reasons | 6 | 5

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I - Donepezil | Arm II - Control | Total
Number analyzed (Participants) | 99 | 99 | 198
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 83 | 155
  >=65 years | 27 | 16 | 43
Age, Continuous [Median (Full Range); unit: years] | 56.1 [19 to 84] | 54.9 [19 to 81] | 55.1 [19 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 50 | 106
  Male | 43 | 49 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 96 | 97 | 193
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 91 | 90 | 181
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 99 | 99 | 198

OUTCOME MEASURES:

1. Primary Outcome: Memory as Quantified by HVLT-immediate Recall
Description: Memory is quantified using the Hopkins Verbal Learning Test (HVLT) - immediate recall. Participants are asked to recall 12 words. Each recalled word is given one point. They are given three trials. The total score is the sum of the recalled words. The range for HVLT-Immediate recall is 0 to 36. Higher scores represent better memory.
Time Frame: 24 weeks
Population: Participants with 24 week HVLT data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I - Donepezil | Arm II - Control
Number analyzed (Participants) | 72 | 73
units on a scale | 22.5 (0.45) | 22.2 (0.45)
Statistical Analysis 1: Comparison: Arm I - Donepezil vs Arm II - Control; Null Hypothesis: No difference in immediate recall memory at 24 weeks; Test type: Superiority or Other; p = .62, Mixed Models Analysis — Not adjusted for multiple comparisons

2. Primary Outcome: Memory as Quantified by the HVLT-discrimination
Description: In the Hopkins Verbal Learning Test - discrimination, participants are given lists of 12 correct words and 12 incorrect words. HVLT-discrimination is the number of correctly recognized words minus the number incorrectly recognized. The range for this outcome measure is -12 to 12. Higher scores represent better memory.
Time Frame: 24 weeks
Population: Number of participants with 24 week memory data
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I - Donepezil | Arm II - Control
Number analyzed (Participants) | 72 | 73
units on a scale | 10.1 (0.24) | 9.2 (0.24)
Statistical Analysis 1: Comparison: Arm I - Donepezil vs Arm II - Control; Null Hypothesis: No difference in discrimination memory between the two groups; Test type: Superiority or Other; p = .007, Mixed Models Analysis — Not adjusted for multiple comparisons

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Analysis includes everyone with post-treatment AE/toxicity data.
Arm/Group | Arm I - Donepezil | Arm II - Control
Serious Adverse Events (participants affected / at risk) | 12/96 | 10/92
Other Adverse Events (participants affected / at risk) | 88/96 | 80/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Donepezil (N=96) | Arm II - Control (N=92)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Auditory/Ear - Other (Ear and labyrinth disorders) | 0 (0) | 1 (3)
Cognitive Disturbance (Psychiatric disorders) | 0 (0) | 1 (2)
Confusion (Nervous system disorders) | 0 (0) | 1 (2)
Death NOS (General disorders) | 1 (1) | 2 (2)
Dental: peridontal disease (General disorders) | 0 (0) | 1 (1)
Dental: teeth (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (5) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hearing (Ear and labyrinth disorders) | 1 (2) | 1 (3)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Mood Alteration: Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Neuropathy: cranial: CN II Vision (Nervous system disorders) | 0 (0) | 1 (3)
Neuropathy: cranial: CN VII Motor-face; Sensory-taste (Nervous system disorders) | 0 (0) | 1 (3)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 1 (1)
Pain - Other (Nervous system disorders) | 1 (1) | 0 (0)
Pain: Back (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (fainting) (General disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Donepezil (N=96) | Arm II - Control (N=92)
Anorexia (Psychiatric disorders) | 21 (33) | 13 (17)
Cognitive Disturbance (Psychiatric disorders) | 26 (64) | 28 (73)
Constipation (Gastrointestinal disorders) | 3 (6) | 5 (11)
Diarrhea (Gastrointestinal disorders) | 24 (29) | 7 (13)
Dizziness (Ear and labyrinth disorders) | 5 (5) | 7 (13)
Fatigue (Metabolism and nutrition disorders) | 55 (105) | 61 (122)
Headache (Nervous system disorders) | 42 (70) | 40 (73)
Insomnia (General disorders) | 43 (81) | 36 (70)
Memory Impairment (Nervous system disorders) | 34 (83) | 34 (91)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (5) | 5 (11)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 32 (58) | 26 (48)
Nausea (Gastrointestinal disorders) | 13 (19) | 17 (21)
Vomiting (Gastrointestinal disorders) | 8 (10) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes